CLINICAL TRIAL: NCT03848104
Title: Evaluation of the Use of Cefoxitin in Combination in Continuous Parenteral Administration in the Treatment of Bone and Joint Infections
Status: Completed | Type: Observational
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Principal Investigator, Eugénie MABRUT, clinical research assistant, Hospices Civils de Lyon
Other Study IDs: 18-079
Record Dates: First submitted 2019-02-19; First posted 2019-02-20 (Actual); Last update posted 2019-02-22 (Actual); Status verified 2019-02

CONDITIONS: Antibiotic Reaction; Bone and Joint Infection
Keywords: cefoxitin; Bone and Joint Infection
MeSH Terms: interventions — Cefoxitin

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- bone and joint infection treated with cefoxitin: patients having had a bone or joint infection treated by cefoxitin in combination. Cefoxitin has been administered by continuous way, at home. A serum dosage of cefoxitin has been systematically achieved at equilibrium.
  Interventions: Other: bone and joint infection treated with cefoxitin

INTERVENTIONS:
Other: bone and joint infection treated with cefoxitin — the patients had cefoxitin in combination in continuous parenteral administration to treat their bone / joint infection

SUMMARY:
Cephamycin related to 2nd generation cephalosporins, the use of cefoxitin has long been limited to antibiotic prophylaxis. Because of its spectrum (sensitive staphylococci, enterobacteria including ESBL, streptococci, anaerobes), its stability and its low cost, it could be useful in curative bone and joint infections, especially in case of infection polymicrobial disease in patients for whom antibiotic alternative per os is limited.

ELIGIBILITY:
Inclusion Criteria:

* patients havind had a bon and joint infeciton treated with cefoxitin in combination in continuous parenteral administration

Exclusion Criteria:

-

Ages: 18 Years to 100 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: patients havind had a bon and joint infeciton treated with cefoxitin in combination in continuous parenteral administration managed at the Croix-Rousse Hospital
Sampling Method: Non-Probability Sample
Enrollment: 35 (Actual)
Dates: Start 2018-01-01 (Actual); Primary Completion 2018-03-01 (Actual); Study Completion 2018-04-01 (Actual)

PRIMARY OUTCOMES:
Rate of Treatment Failure | Outcome is measured at the end of follow-up (usually between 12 and 24 months after antibiotic therapy disruption
  Treatment failure is defined by local clinical and/or microbiological relapse; and/or need for additional surgery; death of septic origin

SECONDARY OUTCOMES:
Rate of use of this strategy | Outcome is measured at the end of follow-up (usually between 12 and 24 months after antibiotic therapy disruption
  Descriptions of patients managed with this strategy

CONTACTS AND LOCATIONS:
Overall Officials: Tristan Ferry, Md,PhD, Principal Investigator — Hospices Civils de Lyon
Locations (1):
- Hospices Civils de Lyon, Lyon, France

IPD SHARING:
Plan to Share IPD: Undecided